CLINICAL TRIAL: NCT04054323
Title: The Efficacy of Physical Activity on Improving Health Outcomes for Renal Transplant Patients and Their Caregivers
Brief Title: The Efficacy of Physical Activity on Improving Health Outcomes for Renal Transplant Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no physical therapist available
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jennifer Steel, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO18080372
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2021-05

CONDITIONS: Chronic Kidney Diseases
Keywords: Exercise; CKD; Graft Survival; Transplant Waitlist
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient Physical Activity Arm (Experimental): Patients only receive physical activity intervention.
  Interventions: Behavioral: Physical Activity Intervention
- Dyadic Physical Activity Arm (Experimental): Patients and caregivers both receive physical activity intervention.
  Interventions: Behavioral: Physical Activity Intervention

INTERVENTIONS:
Behavioral: Physical Activity Intervention — The physical activity intervention will include basic skill training during which the participant will be instructed on the use of (1) the activPAL physical activity device for the tracking of time spent sitting, standing, and walking, (2) tools to monitor exercise intensity, including ratings of perceived exertion, (3) an exercise calendar for setting a specific schedule for the completion of the home exercise program using the exercise videos posted on our website, (4) use of the exercise equipment that will be used in the home program (Therabands), and (5) strategies for reduction of sedentary behavior that target prolonged sitting and encourages frequent activity breaks. Duration of intervention is 6 months.

SUMMARY:
The purpose of this study is to see whether a physical activity intervention improves fitness, strength and reduces sedentary behavior. The investigators are also interested in determining if changes will improve quality of life and outcomes associated with renal transplant waitlist.

DETAILED DESCRIPTION:
Over 30 million people have chronic kidney disease (CKD) and nearly 100,000 people are awaiting renal transplant for end stage renal disease (ESRD). Renal transplant, when compared to dialysis, improves quality of life, is more cost-effective, and reduces the risk of cardiovascular disease. However, many patients who are eligible for transplant become deconditioned while waiting for organ transplantation, and may be taken off the transplant waitlist for concerns the patient will not be able to tolerate surgery. Moreover, poor physical functioning prior to transplant was associated with a 2.5-fold increased risk for delayed graft function and 2.30 fold higher risk of patient death after renal transplant. Our team has also shown that functional limitations, such as slower gait speed and poorer grip strength, were associated with not being waitlisted for transplant and decreased survival in all transplant candidates undergoing evaluation. Functional limitation may reduce the individuals' overall level of physical activity, which can increase further disability. While physical activity (PA) interventions have been shown to be effective in reducing morbidity and mortality in other chronic diseases, no study has tested the efficacy of a PA intervention in patients awaiting renal transplant. Family caregivers are integral in the care of renal transplant candidates. Decades of research has shown that family caregivers are at increased risk for cardiovascular disease (CVD) and mortality when compared to non-caregivers. Investigators propose to include the family caregivers in the PA intervention to improve patient adherence to the intervention while reducing the caregivers' risk for CVD. The proposed study addresses several of the recommendations from consensus meeting on exercise in solid organ transplant which included testing a PA intervention in a large-scale trial with both standard and surrogate markers, using a novel technology-assisted delivery of the intervention, and focusing on mechanisms linking PA with health outcomes.

ELIGIBILITY:
Inclusion criteria

* Patient:

  * Waitlisted for renal transplant
  * =>21 years of age
* Caregiver:

  * Primary caregiver for patient
  * =>21 years of age

Exclusion criteria:

* Patient:

  * Active suicidal ideation
  * Thought disorder
  * Delusions
  * Hallucinations
  * Recent myocardial infarction, heart attack, or stroke
  * Planned elective surgeries for joint replacement
* Caregiver:

  * Active suicidal ideation
  * Thought disorder
  * Delusions
  * Hallucinations
  * Recent myocardial infarction, heart attack, or stroke
  * Planned elective surgeries for joint replacement

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change of Gate Speed from Baseline vs. 6 months | Baseline vs. 6 months
  Measured as meters/second

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | Baseline vs. 6 months
  Metabolic Equivalence of Task (MET) to Access Daily Activity Level
Medical Outcome Survey - Short Form 36 | Baseline vs. 6 months
  Quality of Life Assessment (0 -100)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Steel, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Montefiore Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No